CLINICAL TRIAL: NCT03825224
Title: Evaluation of MyoStrain™ in Clinical Practice
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00142902
Record Dates: First submitted 2019-01-04; First posted 2019-01-31 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Failure; Coronary Artery Disease; Sarcoidosis; Amyloidosis; Lupus; Myocarditis; Drug Toxicity
Keywords: MRI; SENC MyoStrain
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Sarcoidosis; Amyloidosis; Myocarditis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: Diagnostic Test: Myostrain — This test measures the contraction of the heart muscle in one to three heartbeats per plane. It's a pulse sequence that produces images that reveal the underlying contraction fo the muscle of a healthy heart and associated weaknesses in case of disease.

SUMMARY:
Evaluate MyoStrain cardiac MRI pulse sequence in Clinical practice

DETAILED DESCRIPTION:
Evaluate MyoStrain cardiac MRI pulse sequence in Clinical practice to determine how the use may alter treatment decisions and clinical outcomes in patients who are undergoing cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled for diagnostic testing with commercially available imaging modality (cardiac MRI)
* The patient population will include (but not limited to), those being evaluated for heart disease and heart failure that may be related to vascular disease (coronary artery disease), drug related heart failure (chemotherapy, alcohol), inflammatory systemic conditions (sarcoidosis, amyloidosis, lupus), myocarditis, and/or infectious etiologies
* Provided written informed consent

Exclusion Criteria:

* Contraindication to Magnetic Resonance Imaging

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Population will consist of patients scheduled for diagnostic testing with cardiac MRI
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluate workflow for MyoStrain testing | Baseline
  Survey the CMR interpreter to see how Myostrain impacted their interpretation and survey the referring clinician after receiving the CMR report.
  Survey Questions using 5-point Likert and binary reporting scale. The lower numbers represent positive feedback. Example listed below:
  CARDIAC MRI INTERPRETATION QUESTIONS FOR READER (CARDIOLOGIST OR RADIOLOGIST)
  How easy was it to interpret the additional Myostrain sequence information? 1 2 3 4 5
  (1=Very Helpful 2=Helpful 3=Indifferent 4=Unhelpful 5=Very Unhelpful)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Everist, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korosoglou G, Youssef AA, Bilchick KC, Ibrahim el-S, Lardo AC, Lai S, Osman NF. Real-time fast strain-encoded magnetic resonance imaging to evaluate regional myocardial function at 3.0 Tesla: comparison to conventional tagging. J Magn Reson Imaging. 2008 May;27(5):1012-8. doi: 10.1002/jmri.21315. PMID 18407541
- [Background] Sugimori H, Oyama-Manabe N, Ishizaka K, Hamaguchi H, Sakata M. Comparison of SPAMM and SENC methods for evaluating peak circumferential strain at 3T. Magn Reson Med Sci. 2013 Mar 25;12(1):69-75. doi: 10.2463/mrms.2012-0045. Epub 2013 Mar 11. PMID 23474965
- [Background] Ohyama Y, Ambale-Venkatesh B, Chamera E, Shehata ML, Corona-Villalobos CP, Zimmerman SL, Hassoun PM, Bluemke DA, Lima JAC. Comparison of strain measurement from multimodality tissue tracking with strain-encoding MRI and harmonic phase MRI in pulmonary hypertension. Int J Cardiol. 2015 Mar 1;182:342-348. doi: 10.1016/j.ijcard.2015.01.016. Epub 2015 Jan 6. PMID 25590963
- [Background] Altiok E, Neizel M, Tiemann S, Krass V, Becker M, Zwicker C, Koos R, Kelm M, Kraemer N, Schoth F, Marx N, Hoffmann R. Layer-specific analysis of myocardial deformation for assessment of infarct transmurality: comparison of strain-encoded cardiovascular magnetic resonance with 2D speckle tracking echocardiography. Eur Heart J Cardiovasc Imaging. 2013 Jun;14(6):570-8. doi: 10.1093/ehjci/jes229. Epub 2012 Nov 12. PMID 23148082
- [Background] Korosoglou G, Gitsioudis G, Voss A, Lehrke S, Riedle N, Buss SJ, Zugck C, Giannitsis E, Osman NF, Katus HA. Strain-encoded cardiac magnetic resonance during high-dose dobutamine stress testing for the estimation of cardiac outcomes: comparison to clinical parameters and conventional wall motion readings. J Am Coll Cardiol. 2011 Sep 6;58(11):1140-9. doi: 10.1016/j.jacc.2011.03.063. PMID 21884952
- [Background] Korosoglou G, Lehrke S, Wochele A, Hoerig B, Lossnitzer D, Steen H, Giannitsis E, Osman NF, Katus HA. Strain-encoded CMR for the detection of inducible ischemia during intermediate stress. JACC Cardiovasc Imaging. 2010 Apr;3(4):361-71. doi: 10.1016/j.jcmg.2009.11.015. PMID 20394897
- [Background] Korosoglou G, Lossnitzer D, Schellberg D, Lewien A, Wochele A, Schaeufele T, Neizel M, Steen H, Giannitsis E, Katus HA, Osman NF. Strain-encoded cardiac MRI as an adjunct for dobutamine stress testing: incremental value to conventional wall motion analysis. Circ Cardiovasc Imaging. 2009 Mar;2(2):132-40. doi: 10.1161/CIRCIMAGING.108.790105. Epub 2009 Jan 26. PMID 19808579
- [Background] Korosoglou G, Futterer S, Humpert PM, Riedle N, Lossnitzer D, Hoerig B, Steen H, Giannitsis E, Osman NF, Katus HA. Strain-encoded cardiac MR during high-dose dobutamine stress testing: comparison to cine imaging and to myocardial tagging. J Magn Reson Imaging. 2009 May;29(5):1053-61. doi: 10.1002/jmri.21759. PMID 19388131
- [Background] Korosoglou G, Giusca S, Gitsioudis G, Erbel C, Katus HA. Cardiac magnetic resonance and computed tomography angiography for clinical imaging of stable coronary artery disease. Diagnostic classification and risk stratification. Front Physiol. 2014 Aug 6;5:291. doi: 10.3389/fphys.2014.00291. eCollection 2014. PMID 25147526
- [Background] Neizel M, Korosoglou G, Lossnitzer D, Kuhl H, Hoffmann R, Ocklenburg C, Giannitsis E, Osman NF, Katus HA, Steen H. Impact of systolic and diastolic deformation indexes assessed by strain-encoded imaging to predict persistent severe myocardial dysfunction in patients after acute myocardial infarction at follow-up. J Am Coll Cardiol. 2010 Sep 21;56(13):1056-62. doi: 10.1016/j.jacc.2010.02.070. PMID 20846606
- [Background] Neizel M, Lossnitzer D, Korosoglou G, Schaufele T, Peykarjou H, Steen H, Ocklenburg C, Giannitsis E, Katus HA, Osman NF. Strain-encoded MRI for evaluation of left ventricular function and transmurality in acute myocardial infarction. Circ Cardiovasc Imaging. 2009 Mar;2(2):116-22. doi: 10.1161/CIRCIMAGING.108.789032. Epub 2009 Jan 26. PMID 19808577
- [Background] Koos R, Altiok E, Doetsch J, Neizel M, Krombach G, Marx N, Hoffmann R. Layer-specific strain-encoded MRI for the evaluation of left ventricular function and infarct transmurality in patients with chronic coronary artery disease. Int J Cardiol. 2013 Jun 5;166(1):85-9. doi: 10.1016/j.ijcard.2011.10.004. Epub 2011 Nov 8. PMID 22071039
- [Background] Oyama-Manabe N, Ishimori N, Sugimori H, Van Cauteren M, Kudo K, Manabe O, Okuaki T, Kamishima T, Ito YM, Tsutsui H, Tha KK, Terae S, Shirato H. Identification and further differentiation of subendocardial and transmural myocardial infarction by fast strain-encoded (SENC) magnetic resonance imaging at 3.0 Tesla. Eur Radiol. 2011 Nov;21(11):2362-8. doi: 10.1007/s00330-011-2177-4. Epub 2011 Jun 18. PMID 21688005
- [Background] Youssef A, Ibrahim el-SH, Korosoglou G, Abraham MR, Weiss RG, Osman NF. Strain-encoding cardiovascular magnetic resonance for assessment of right-ventricular regional function. J Cardiovasc Magn Reson. 2008 Jul 4;10(1):33. doi: 10.1186/1532-429X-10-33. PMID 18601713
- [Background] Shehata ML, Basha TA, Tantawy WH, Lima JA, Vogel-Claussen J, Bluemke DA, Hassoun PM, Osman NF. Real-time single-heartbeat fast strain-encoded imaging of right ventricular regional function: normal versus chronic pulmonary hypertension. Magn Reson Med. 2010 Jul;64(1):98-106. doi: 10.1002/mrm.22408. PMID 20572146
- [Background] Hamdan A, Thouet T, Kelle S, Paetsch I, Gebker R, Wellnhofer E, Schnackenburg B, Fahmy AS, Osman NF, Fleck E. Regional right ventricular function and timing of contraction in healthy volunteers evaluated by strain-encoded MRI. J Magn Reson Imaging. 2008 Dec;28(6):1379-85. doi: 10.1002/jmri.21526. PMID 19025945
- [Background] Hamdan A, Thouet T, Kelle S, Wellnhofer E, Paetsch I, Gebker R, Schnackenburg B, Fahmy AS, Osman NF, Bornstedt A, Fleck E. Strain-encoded MRI to evaluate normal left ventricular function and timing of contraction at 3.0 Tesla. J Magn Reson Imaging. 2009 Apr;29(4):799-808. doi: 10.1002/jmri.21684. PMID 19306402
- [Background] Freed BH, Tsang W, Bhave NM, Patel AR, Weinert L, Yamat M, Vicedo BM, Dill K, Mor-Avi V, Gomberg-Maitland M, Lang RM. Right ventricular strain in pulmonary arterial hypertension: a 2D echocardiography and cardiac magnetic resonance study. Echocardiography. 2015 Feb;32(2):257-63. doi: 10.1111/echo.12662. Epub 2014 Jun 28. PMID 24975738

DOCUMENTS (1):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT03825224/Prot_000.pdf